## REFINING AND PILOTING A TEXT MESSAGING INTERVENTION TO DELAY ALCOHOL INITIATION AND REDUCE ALCOHOL USE ESCALATION AMONG ABSTAINER AND LIGHTER DRINKER COLLEGE STUDENTS

NCT03750838 11/16/2023

## **Analytic Plan**

To assess feasibility of the intervention, we examined targeted recruitment, enrollment, and retention rates. To feasibility, we examined response rates for text message intervention rating for those assigned to the intervention condition. For acceptability, we assessed overall ratings of acceptability as well as mean ratings of content area-specific text messages. Rates of alcohol initation (yes/no) were examined at each time point as were means and standard deviations of the number of drinks per week at each time point.